CLINICAL TRIAL: NCT07234799
Title: Feasibility Testing of a Dyadic Exercise Program for Patients Undergoing Thoracic Radiotherapy and Their Family Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0744; NCI-2025-07868 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-10-22; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Protocol (Experimental): The protocol will be comprised of up to 15 exercise sessions over the course of participants' 5-6 weeks radiation treatment period with each session lasting up to 60 minutes. Exercise sessions are a combination of resistance, aerobic, and flexibility training using bodyweight and/or elastic bands for resistance.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Study participants will engage in 7-10 exercises per session targeting major muscle groups (e.g. quadriceps, hamstrings, glutes, back, chest, arms, abdominal muscles). Movements will alternate between the lower and upper body thus allowing ample time for muscle-group recovery between exercises.

SUMMARY:
The goal of this study is to examine the feasibility and acceptability of an exercise intervention for patients undergoing thoracic radiation and their family caregivers.

DETAILED DESCRIPTION:
Primary Objectives:

1. Examine the feasibility and acceptability of an exercise program
2. Examine an initial sign for intervention efficacy by examining pre/post-test scores for patients' objective physical function and patient and caregiver subjective physical and mental quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with a non-small cell lung cancer or esophageal cancer and going to receive at least 24 fractions thoracic RT
* Have an ECOG performance status of ≤2
* Have a family caregiver (e.g., spouse, sibling, adult child) willing and able (self-identified) to participate in the exercise program

Both patient and caregiver must meet all the following criteria:

* Be ≥18 years old
* Be able to read and speak English
* Be able to provide informed consent

Exclusion Criteria:

* A patient who meets the following criteria will be excluded from participating in this study:
* Cognitive deficits noted in the medical records and/or cognitive deficits that would impede the completion of self-report instruments as deemed by the patient's attending radiation oncologist.
* Experiences contraindications to exercise as determined by the clinical team
* Regularly (self-defined) participates in an exercise program in the year prior to diagnosis

A patient and caregiver who is pregnant (medical notes and/or self-identified, respectively) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2028-05-04 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | Through study completion; an average of 1 year
  Patients and caregivers will complete the Medical Outcomes. Study 36-item short-form survey (SF-36) assessing 8 distinct domains of QOL

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, MA,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org